CLINICAL TRIAL: NCT02305797
Title: A Randomized Double-Blind, Placebo Controlled, Flexible Dose, Parallel Group Study of Extended-Release Lorazepam (EDG004) for the Treatment of Generalized Anxiety Disorder (GAD)
Brief Title: EDG004 Treatment of Adult Patients With Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Edgemont Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDG004-003
Record Dates: First submitted 2014-11-25; First posted 2014-12-03 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2016-07

CONDITIONS: Generalized Anxiety Disorder (GAD)
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EDG004 (Experimental): EDG004 - Extended release lorazepam capsules
  Interventions: Drug: Extended-release lorazepam
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended-release lorazepam — Extended-release lorazepam capsules
  Other Names: EDG004
  Arms: EDG004
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of EDG004 compared to placebo for the treatment of adult patients with GAD, diagnosed by Diagnostic and Statistical Manual of Mental Disorders, 5th Ed. (DSM-5) and confirmed by the Mini International Neuropsychiatric Interview (MINI 7.0). Efficacy will be measured by a statistically significant greater mean reduction from baseline compared to endpoint in anxiety symptoms as measured by the total score of the clinician-rated Hamilton Rating Scale for Anxiety (HAM-A) for the EDG004 treatment group compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-65 years and
* Diagnosed with GAD and
* No other psychiatric conditions, and are otherwise medically healthy.

Exclusion Criteria:

* Women who are pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Investigational Sites, Multiple Locations, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 44 centers in the United States.
Pre-assignment Details: Patients were evaluated for eligibility during a screening period and underwent a washout from prior and concomitant medications using protocol-specified guidelines, where applicable.
Groups:
- EDG004: EDG004
  EDG004: EDG004
  Extended release lorazepam capsules dosed once daily at 1, 2, 3, 4, 5, or 6 mg/day.
- Placebo: Placebo
  Placebo: Placebo
Period: Overall Study
Arm/Group | EDG004 | Placebo
Started | 247 | 248
Completed | 202 | 210
Not Completed | 45 | 38
Not completed — Adverse Event | 11 | 2
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Lack of Efficacy | 6 | 0
Not completed — Lost to Follow-up | 5 | 11
Not completed — Pregnancy | 0 | 2
Not completed — Noncompliance | 14 | 12
Not completed — Reason not collected | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 495 patients were randomly assigned to a treatment group and received at least one dose of study treatment. The mITT Set included 239 patients randomly assigned to EDG004 and 240 patients randomly assigned to placebo.
Groups:
- EDG004: EDG004
  EDG004: EDG004
- Total: Total of all reporting groups
Arm/Group | EDG004 | Placebo | Total
Number analyzed (Participants) | 239 | 240 | 479
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.36) | 35.9 (11.96) | 36.2 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 70 | 138
  Male | 171 | 170 | 341
Region of Enrollment [Number; unit: participants]
  United States | 239 | 240 | 479

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at Visit 7 (Day 42)
Description: HAM-A Total Score was rated by the clinician. Scores range from 0 to 56. A lower score is favorable. Baseline was defined as the last non-missing value prior to receiving double-blind study drug.
Time Frame: Day 42 (Visit 7)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | EDG004 | Placebo
Number analyzed (Participants) | 239 | 240
Score on scale | -9.01 (0.47) | -8.93 (0.48)

2. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity (CGI-S) Score at Visit 7 (Day 42)
Description: Measured on a 7-point scale 1 = Normal, not at all ill; 2 = Borderline mentally ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill. Baseline was defined as the last non-missing value prior to receiving double-blind study drug.
Time Frame: Day 42 (Visit 7)
Population: The modified Intent-to-treat (mITT) population was used for all analyses.
Measure: Least Squares Mean (Standard Error); unit: CGI-S score
Arm/Group | EDG004 | Placebo
Number analyzed (Participants) | 239 | 240
CGI-S score | -1.14 (0.072) | -1.10 (0.071)

ADVERSE EVENTS:
Arm/Group | EDG004 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/247 | 0/248
Other Adverse Events (participants affected / at risk) | 131/247 | 64/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDG004 (N=247) | Placebo (N=248)
Intentional Self-Injury (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDG004 (N=247) | Placebo (N=248)
Nausea (Gastrointestinal disorders) | 18 (21) | 13 (15)
Fatigue (General disorders) | 32 (36) | 7 (7)
Headache (Nervous system disorders) | 16 (19) | 19 (26)
Dizziness (Nervous system disorders) | 23 (23) | 9 (10)
Somnolence (Nervous system disorders) | 42 (50) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No